CLINICAL TRIAL: NCT03029689
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Effect of Raltegravir Intensification (1.200 mg QD) on the Gut Microbiota of Chronically HIV-1 Infected Subject Over Time: THE RAGTIME
Brief Title: Clinical Trial to Evaluate the Effect of Raltegravir Intensification (1.200 mg QD) on the Gut Microbiota of Chronically HIV-1 Infected Subject Over Time: THE RAGTIME STUDY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RAGTIME
Record Dates: First submitted 2017-01-11; First posted 2017-01-24 (Estimated); Results first posted 2025-04-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: HIV
Keywords: HIV infection; Gut microbiome; Raltegravir; Raltegravir intensification; Bacterial richness
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current ART + Raltegravir (Experimental): Current ART + Raltegravir
  Interventions: Drug: Raltegravir; Drug: Current ART
- Current ART + placebo (Placebo Comparator): Current ART + placebo
  Interventions: Drug: Placebo; Drug: Current ART

INTERVENTIONS:
Drug: Raltegravir — Raltegravir 1200 mg (2 tablets x 600mg) once daily plus current ART during 48 weeks from randomization
  Other Names: NP
  Arms: Current ART + Raltegravir
Drug: Placebo — Placebo (2 tablets of placebo) once daily plus current ART during 48 weeks from randomization.
  Other Names: NP
  Arms: Current ART + placebo
Drug: Current ART — 3-drug antiretroviral treatment including PI/r/c or NNRTI
  Other Names: NP

SUMMARY:
The project presented here will be the first prospective, randomized evaluation of the effect of ART on the structure and function of the gut microbiome. This study provides a unique opportunity to understand the benefits of ART with high intestinal penetration on the gut microbiome. It is thus a key study to understand the bidirectional interactions between the microbiome and the host in people living with HIV/AIDS.

DETAILED DESCRIPTION:
The gut microbiome is essential for the maturation of the neonatal immune system and the adequate development and function of adult immune responses. HIV-1 infection in children and adults exerts a rapid and severe depletion of gut-associated lymphoid tissue, which damages the intestinal barrier, allowing translocation of gut commensal bacteria into the systemic circulation. Bacterial translocation causes chronic inflammation and immune activation, which lead to immune deterioration and premature aging of HIV-1-infected subjects, including metabolic disturbances, cardiovascular diseases, cognitive disorders and HIV-associated cancers. Persistence of residual HIV-1 replication in the presence of ART has been associated to incomplete HIV-1 suppression in gut lymphatic tissues due to suboptimal tissular penetration of PI/s or NNRTIs.

In previous work in our institute, the investigators have observed that HIV-1 infection is independently associated with significant reductions in the gut microbiome richness, which is, in turn, are inversely correlated with systemic inflammation. Reduced microbial richness, for example, has been associated with intestinal inflammatory diseases and well as with metabolic syndrome, diabetes and obesity and correlated with metabolic markers.

Recovering bacterial richness might thus have a positive impact on immune activation, chronic inflammation and the overall health of HIV-infected individuals. However, achieving that goal will possibly require, alongside potential bacterial supplementations, the use of ART with high penetration into gut lymphoid tissue to limit as much as possible the continued damage exerted by residual HIV replication on the GALT. Antiretroviral drugs with higher intestinal penetration like raltegravir may be more effective at recovering the intestinal microbiome composition and function than those with lower gut penetration like darunavir or the NNRTIs. Thereby, raltegravir intensification could be associated with increases in intestinal microbial richness, implying an improvement on intestinal and overall health.

Despite the lack of evidence on that regard, previous studies from our group and others would favor that hypothesis. Residual HIV-1 replication in plasma can be deterred by ART intensification with raltegravir, which is, in part, due to the high penetration of raltegravir in intestinal tissues. Moreover, raltegravir intensification decreases peripheral CD8 T-cell activation CD45RA (-) and creates a transient CD4 T-cell redistribution, which revert after raltegravir withdrawal.

The project presented here will be the first prospective, randomized evaluation of the effect of ART on the structure and function of the gut microbiome. This study provides a unique opportunity to understand the benefits of ART with high intestinal penetration on the gut microbiome. It is thus a key study to understand the bidirectional interactions between the microbiome and the host in people living with HIV/AIDS

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Documented HIV infection
3. Stable 3-drug antiretroviral treatment including PI/r/c or NNRTI for at least 6 months.
4. Plasma HIV-1 RNA load <50 copies/mL for at least 12 months.
5. Signed Informed Consent

Exclusion Criteria:

1. PI/r monotherapy
2. INSTI therapy during the previous 6 months
3. Evidence of previous INSTI resistance
4. Creatine clearance <50 mL/min
5. Child- Pugh B or C
6. History of active uncontrolled GI disorders or diseases including:

   6.1. Major surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the previous 5 years.

   6.2. Any major bowel resection at any time.

   6.3. Any chronic digestive disease such as peptic ulcer, Crohn's disease, ulcerative colitis, coeliac disease, confirmed intolerance to lactose or indeterminate colitis.

   6.4. Persistent infectious gastroenteritis, colitis or gastritis; persistent or chronic diarrhea of unknown etiology; Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated)

   6.5. Irritable bowel syndrome (moderate-severe)

   6.6. Chronic constipation

   6.7. Active proctitis
7. Antibiotic therapy within the previous 2 months
8. In women, pregnancy or breastfeeding*.

   * Female subjects of childbearing potential must not be pregnant, not be planning a pregnancy or breast-feeding. Sexually active women must be willing to use two approved methods of contraception (including condoms, diaphragm, spermicides, hormonal methods and/or intrauterine devices) from baseline until the end of the clinical trial. Sexually active men in heterosexual relationships must be willing to use two approved method of contraception with their partners from baseline until the end of the clinical trial.
   * condom use is considered as an additional method of contraception only and cannot be the only method of contraception used as not been considered an effective method by the Clinical Trial Facilitation Group (CTFG) guidelines.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Current ART + Raltegravir | Current ART + Placebo
Started | 40 | 21
Completed | 37 | 17
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Current ART + Raltegravir | Current ART + Placebo | Total
Number analyzed (Participants) | 37 | 17 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 16 | 52
  >=65 years | 1 | 1 | 2
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [38 to 56] | 52 [47 to 58] | 52 [41 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 32 | 16 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 21 | 6 | 27
  Unknown or Not Reported | 14 | 9 | 23
Region of Enrollment [Number; unit: participants]
  Spain | 37 | 17 | 54

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Gene Richness (Observed Unique Genes). Analysis of the Composition, Structure and Function of the Intestinal Microbiome. *
Description: -* Structure and composition of the microbiome. DNA will be extracted and purified from fecal samples and cryopreserved at -80ºC until amplification. The purified DNA will be amplified using Illumina-tagged primers to amplify the V3 and V4 16S ribosomal DNA (rDNA) regions. PCR reactions will be performed in triplicate to preserve diversity. Pooled triplicates will be sequenced ensuring adequate sampling depth.
  -Function of the bacteriome. The gene content will be inferred from the abundance of each bacteria in the intestinal bacteriome according to the 16S rDNA information
Time Frame: From baseline to 48 weeks
Measure: Median (Inter-Quartile Range); unit: Number of unique genes detected
Arm/Group | Current ART + Raltegravir | Current ART + Placebo
Number analyzed (Participants) | 37 | 17
Number of unique genes detected
  Gene richness at baseline | 768358 [663708 to 879113] | 730732 [552699 to 869340]
  Gene richness at timepoint 12 | 767756 [600703 to 834276] | 808911 [721094 to 832215]
  Gene richness at timepoint 24 | 724452 [605639 to 825037] | 777452 [695461 to 872279]
  Gene richness at timepoint 48 | 718824 [624788 to 848524] | 860913 [745053 to 882858]

2. Secondary Outcome: Association of the Gut Microbiome With Inflammation Markers
Description: IL-6, IP-10
Time Frame: From baseline to week 48
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Current ART + Raltegravir | Current ART + Placebo
Number analyzed (Participants) | 37 | 17
pg/ml
  IL-6 at baseline | 1.32 [1.14 to 1.78] | 1.53 [1.41 to 1.78]
  IL-6 at week 12 | 1.52 [1.09 to 1.81] | 1.48 [1.23 to 1.67]
  IL-6 at week 24 | 1.25 [1.06 to 1.65] | 1.38 [1.14 to 1.58]
  IL-6 at week 48 | 1.28 [1.13 to 1.58] | 1.3 [1.1 to 1.51]
  IP-10 at baseline | 102.99 [84.95 to 126.16] | 97.44 [80.65 to 123.53]
  IP-10 at week 12 | 104.7 [84.7 to 125.17] | 108.6 [79.13 to 127.13]
  IP-10 at week 24 | 104.6 [81.04 to 122.69] | 99.58 [81.34 to 128.9]
  IP-10 at week 48 | 106.43 [86.79 to 137.85] | 108.55 [85.09 to 118.36]

3. Secondary Outcome: Association of the Gut Microbiome With Coagulation
Description: D-Dimer
Time Frame: From baseline to 48 weeks
Measure: Median (Inter-Quartile Range); unit: ug/ml
Arm/Group | Current ART + Raltegravir | Current ART + Placebo
Number analyzed (Participants) | 37 | 17
ug/ml
  D-Dimer at baseline | 1.99 [1.77 to 2.41] | 2.1 [1.91 to 2.89]
  D-Dimer at week 12 | 2.155 [1.85 to 2.77] | 2.19 [2.03 to 2.45]
  D-Dimer at week 24 | 2.14 [1.69 to 2.47] | 2.22 [1.79 to 2.5]
  D-Dimer at week 48 | 2.22 [1.89 to 2.73] | 2.18 [1.81 to 2.66]

4. Secondary Outcome: Association of the Gut Microbiome With Enterocyte Damage
Description: Intestinal Fatty Acid Binding Protein (I-FABP)
Time Frame: From baseline to 48 weeks
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Current ART + Raltegravir | Current ART + Placebo
Number analyzed (Participants) | 37 | 17
ng/ml
  IFABP at baseline | 0.92 [0.68 to 1.33] | 0.69 [0.6 to 0.89]
  IFABP at week 12 | 0.94 [0.57 to 1.43] | 0.82 [0.65 to 1.19]
  IFABP at week 24 | 1.04 [0.72 to 1.39] | 0.76 [0.65 to 0.98]
  IFABP at week 48 | 0.81 [0.64 to 1.26] | 1.06 [0.75 to 1.13]

5. Secondary Outcome: Association of the Gut Microbiome With Bacterial Translocation and Monocyte Activation
Description: LPS-binding protein (LBP), soluble CD14
Time Frame: From baseline to 48 weeks
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Current ART + Raltegravir | Current ART + Placebo
Number analyzed (Participants) | 37 | 17
ng/ml
  LBP at baseline | 4238 [3395 to 4537] | 4274 [3664 to 5056]
  LBP at week 12 | 4478 [3387 to 4991] | 4313 [3047 to 4792]
  LBP at week 24 | 3879 [3443 to 4839] | 4221 [3467 to 4414]
  LBP at week 48 | 4172 [3649 to 4637] | 4203 [3316 to 4946]
  sCD14 at baseline | 2.41 [2.18 to 2.69] | 2.63 [2.38 to 2.75]
  sCD14 at week 12 | 2.5 [2.26 to 2.6] | 2.61 [2.33 to 2.85]
  sCD14 at week 24 | 2.36 [2.2 to 2.79] | 2.62 [2.35 to 2.73]
  sCD14 at week 48 | 2.48 [2.36 to 2.85] | 2.5 [2.4 to 2.99]

6. Secondary Outcome: Mean Fluorescence Intensity (MFI) Measure of Maturation, Activation, Exhaustion and Immune Senescence Markers in CD4+ and CD8+ T-cells
Description: CCR7, CD28, CD27, HLA-DR, CD38, PD-1, CD57
Time Frame: Differences at week 48
Measure: Median (Inter-Quartile Range); unit: MFI
Arm/Group | Current ART + Raltegravir | Current ART + Placebo
Number analyzed (Participants) | 37 | 17
MFI
  CD28 | 8051 [1471 to 12096] | 8076 [1624 to 12144]
  CD27 | 26002 [676 to 46096] | 27604 [1306 to 47312]
  HLA-DR | 954 [540 to 1955] | 990 [566 to 2244]
  CD38 | 165 [-23.1 to 552] | 130 [-55.6 to 443]
  PD-1 | 1074 [550 to 2086] | 1246 [659 to 2432]
  CD57 | 239 [83.4 to 525] | 226 [75.6 to 524]

7. Secondary Outcome: Association of the Gut Microbiome Composition and Richness With CD4 and CD8+ Counts.
Description: CD4 and CD8+ counts
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: cells/mm^3 of blood
Arm/Group | Current ART + Raltegravir | Current ART + Placebo
Number analyzed (Participants) | 37 | 17
cells/mm^3 of blood
  CD4+ | 696 [554 to 918] | 664 [430 to 658]
  CD8+ | 787 [586 to 968] | 668 [470 to 807]

8. Secondary Outcome: Other Estimators of Richness and Diversity
Description: Shannon
Time Frame: From baseline to 48 weeks
Population: The Shannon Diversity Index (SDI), also known as Shannon-Weaver or Shannon-Wiener Index, is a commonly used metric in ecology and microbiome research to quantify microbial diversity within a sample (alpha diversity). It takes into account both richness (the number of different species and evenness (the relative abundance distribution of species). Higher SDI values reflect greater microbial diversity, while lower SDI values may indicate dysbiosis or a disrupted microbial community.
Measure: Median (Inter-Quartile Range); unit: Shannon index
Arm/Group | Current ART + Raltegravir | Current ART + Placebo
Number analyzed (Participants) | 37 | 17
Shannon index
  Shannon at baseline | 2.90 [2.45 to 3.16] | 2.56 [1.86 to 3.08]
  Shannon at week 12 | 2.91 [2.31 to 3.07] | 2.89 [2.64 to 3.07]
  Shannon at week 24 | 2.65 [2.23 to 3] | 2.56 [2.12 to 2.92]
  Shannon at week 48 | 2.63 [2.13 to 3.10] | 2.97 [2.69 to 3.32]

9. Secondary Outcome: Association of the Gut Microbiome Composition and Richness With CD4/CD8+ Cell Ratio.
Description: CD4/CD8+ cell ratio
Time Frame: Baseline
Population: CD4+/CD8+ ratio
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Current ART + Raltegravir | Current ART + Placebo
Number analyzed (Participants) | 37 | 17
Ratio | 1.10 [0.74 to 1.26] | 0.91 [0.82 to 1.62]

ADVERSE EVENTS:
Time Frame: From baseline to week 48
Arm/Group | Current ART + Raltegravir | Current ART + Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/17
Other Adverse Events (participants affected / at risk) | 1/38 | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Current ART + Raltegravir (N=38) | Current ART + Placebo (N=18)
Adverse event not related to the treatment (Investigations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT03029689/Prot_SAP_000.pdf